CLINICAL TRIAL: NCT02725073
Title: Photodynamic Therapy Using a Novel Photosensitizer in Locally Advanced Hilar Cholangiocarcinoma
Brief Title: Photodynamic Therapy in Locally Advanced Hilar Cholangiocarcinoma
Acronym: PDT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Do Hyun Park, Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERCP-PDT
Record Dates: First submitted 2016-03-20; First posted 2016-03-31 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Treatment Response; Adverse Events; Feasibility
MeSH Terms: interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- photodynamic therapy (Experimental): Photodynamic therapy with a novel photosensitizer and flexible laser catheter
  Interventions: Procedure: Photodynamic therapy

INTERVENTIONS:
Procedure: Photodynamic therapy — Photolon (Belmedpreparaty, Minsk, Republic of Belarus), was administered intravenously at a dose of 2.5 mg/kg at 3 hours before illumination. After advancing a catheter (7 F inner sheath of a plastic stent delivery catheter [MAJ-1419; Olympus America, Center Valley, Pa., USA]) across the biliary stricture using a 0.035-in guidewire, the cylindrical diffuser is inserted into a catheter at the level of the stricture to be treated. Photoactivation (660 nm with a light dose of 100-150J/cm2, and fluence of 0.8-1W/cm2; UPL- FDT; LEMT Research & Development Private Unitary Enterprise, Minsk, Republic of Belarus) is performed

SUMMARY:
To determine the safety and efficacy of photodynamic therapy with a novel photosensitizer and a flexible laser probe in locally advanced hilar cholangiocarcinoma.

DETAILED DESCRIPTION:
Photodynamic therapy (PDT) is a way of producing tissue necrosis with light after prior administration of a photosensitizing agent. The most important advantages include the possibility of combining PDT with other target therapies and repeat the process as needed with a favorable outcomes. The combination of diverse therapeutic modalities is one of the new strategies to enhance oncologic treatments for pancreatic cancer. In order to overcome the limitations of each treatment modalities and to prevent the development of resistance, the application of PDT combined with target therapies, without increasing the toxicity for the patient, is being widely investigated.

PDT has been only extensively studied for the treatment of various superficial skin cancers in the Europe but not available in the United States and Japan due to the overlapping treatment fields. In Korea, the use of first-generation and second-generation photosensitizers are part of the study of Gastroenterology, Dermatology, Otolaryngology, and Gynecology.

Recently, although the investigators have introduced PDT using novel photosensitizers has not yet been used for the treatment of pancreatic cancers. This study aim to determine the safety and efficacy of photodynamic therapy with a novel photosensitizer in locally advanced hilar cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced cholangiocarcinoma confirmed to be unsuitable for surgical resection
2. Exhibiting disease progression without distant metastasis after conventional chemoradiation therapy at multidisciplinary team discussion in Asan Medical Center
3. Pathologically proven cholangiocarcinoma
4. have a negative pregnancy test if appropriate
5. ECOG(Eastern Cooperative Oncology Group) Score 0-2
6. patients to give informed consent and age more than >19 years

Exclusion Criteria:

1. age less than 18 years
2. previous history of PDT
3. uncorrectable coagulopathy
4. refuse to participate
5. pregnancy
6. recent participation in another clinical research trial within 30 days
7. presence of porphyria or hypersensitivity to photosensitizer
8. Creatinine clearance < 45ml

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Treatment response using the Response Evaluation Criteria in Solid Tumours (RECIST) criteria | within 1 month
  Response Evaluation Criteria in Solid Tumours (RECIST) criteria

SECONDARY OUTCOMES:
Adverse events and overall survival | within 1 week
  any procedural adverse events and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Do Hyun Park, Md, PhD, Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Do Hyun Park, Seoul

IPD SHARING:
Plan to Share IPD: Yes